CLINICAL TRIAL: NCT07041216
Title: The Effect of Squishy Toy Squeezing and Palpation Techniques on Peripheral Intravenous Catheter Insertion Success in Pediatric Hematology and Oncology: A Randomized Controlled Trial
Brief Title: Squishy Toy and Palpation in Pediatric IV Success
Acronym: Intravenous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Meltem Gürcan, Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AkdenizUn
Record Dates: First submitted 2025-06-12; First posted 2025-06-27 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pediatric ALL
Keywords: Squishy Toy Squeezing; Peripheral Intravenous Catheter Insertion Success; Palpation Techniques; Pediatric Hematology and Oncology
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Squishy Toy Group (Experimental): In the intervention group, vein suitability was checked using the DIVA score. A tourniquet was applied, the area was cleaned with antiseptic, and the child squeezed a squishy toy 10 times. Afterward, the child stopped using the toy. Once the vein was visible, the catheter was inserted and the tourniquet removed.
  Interventions: Other: Squishy Toy Squeezing
- Palpation Group (Experimental): In this group, once the vein was identified, the area was gently tapped 8 to 10 times using the inner surfaces of four fingers to stimulate blood flow and enhance vein visibility. This light palpation helped increase local circulation, making the vein easier to access. After the palpation procedure, the area was thoroughly cleaned with an antiseptic solution. Once the skin was completely dry, the catheter was inserted under sterile conditions.
  Interventions: Other: Palpation
- Control Group (Other): This group received standard IV insertion with no extra techniques applied.
  Interventions: Other: Routine medical care

INTERVENTIONS:
Other: Squishy Toy Squeezing — In the intervention group, vein suitability was checked using the DIVA score. A tourniquet was applied, the area was cleaned with antiseptic, and the child squeezed a squishy toy 10 times. Afterward,
  Arms: Squishy Toy Group
Other: Palpation — In this group, once the vein was identified, the area was gently tapped 8 to 10 times using the inner surfaces of four fingers to stimulate blood flow and enhance vein visibility. This light palpation helped increase local circulation, making the vein easier to access. After the tapping procedure, the area was thoroughly cleaned with an antiseptic solution. Once the skin was completely dry, the catheter was inserted under sterile conditions.
  Arms: Palpation Group
Other: Routine medical care — This group received standard IV insertion with no extra techniques applied.
  Arms: Control Group

SUMMARY:
This randomized controlled trial investigates the effects of two non-pharmacological techniques-squishy toy squeezing and vein palpation-on the success rate of peripheral intravenous catheter (PIVC) insertion in pediatric hematology and oncology patients. Data collection takes place in the procedure room of a pediatric outpatient clinic. The study includes children who have a Difficult Intravenous Access (DIVA) score of 4 or higher, indicating difficult venous access. Participants are randomly assigned to one of three groups: the squishy toy group, the palpation group, or the control group, which receives standard care.

In the squishy toy group, children use soft, elastic toys to activate hand muscles and improve blood flow, aiming to enhance vein visibility. In the palpation group, the target vein is gently tapped to increase local blood circulation and make the vein more prominent. The control group undergoes catheter insertion without any additional stimulation techniques. All data are recorded using structured forms that collect demographic, clinical, and procedural information. The study aims to determine whether these simple and cost-effective interventions improve the success rate of PIVC insertion in children with difficult venous access.

ELIGIBILITY:
Inclusion Criteria:

* Children identified by the healthcare team as needing peripheral intravenous catheter placement who also have a Difficult Intravenous Access (DIVA) score of 4 or above.

Exclusion Criteria:

* Children unable to squeeze a toy due to physical limitations were excluded from the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Number of IV attempts to successful acces | During the procedure
  During the procedure, the number of intravenous catheter insertion attempts is measured using the catheter documentation form.
Time to successful acces | During the procedure
  During the procedure, the total procedure time is measured using the catheter documentation form.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurcan M, Say B, Yayla N, Atay Turan S. Effectiveness of toy-mediated hand squeezing or palpation in peripheral IV catheterization among pediatric hematology and oncology patients: A randomized controlled trial. Eur J Oncol Nurs. 2025 Dec;79:103005. doi: 10.1016/j.ejon.2025.103005. Epub 2025 Oct 13. PMID 41166835